CLINICAL TRIAL: NCT01173484
Title: Idiopathic Gastroparesis Registry to Define Severity, Treatment Response, and Prognosis Using a Predominant-Symptom Classification
Brief Title: Idiopathic Gastroparesis Registry Using a Predominant-Symptom Classification
Status: Terminated | Type: Observational
Why Stopped: Principal investigator has left the Institution
Sponsor: University of Louisville (Other)
Responsible Party: Sponsor
Other Study IDs: 09-0569
Record Dates: First submitted 2010-07-29; First posted 2010-08-02 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Gastroparesis
Keywords: Idiopathic gastroparesis; Vomiting; Dyspepsia; GERD
MeSH Terms: conditions — Gastroparesis; Vomiting; Dyspepsia; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Vomiting-predominant idiopathic gastroparesis: Vomiting with retching and nausea are the most bothersome symptoms
- Dyspepsia-predominant idiopathic gastroparesis: Unpleasant or troublesome sensation (discomfort or pain) centered in the upper abdomen is the most bothersome symptom; this sensation may be characterized by or associated with upper abdominal fullness, fullness after small meals, bloating, or nausea
- Regurgitation-predominant idiopathic gastroparesis: Effortless regurgitation of acid or undigested food or heartburn is the most bothersome symptom

SUMMARY:
The diagnosis of "gastroparesis" suggests that delayed gastric emptying is the underlying cause of symptoms, but this description fails to explain the variable presentation. There are fundamental differences in causes, symptoms, and prognosis among patients with idiopathic gastroparesis. Understanding these differences is necessary in order to provide effective treatment in these patients. We believe our classification for gastroparesis is a useful tool in the management of patients with idiopathic gastroparesis to predict clinical severity, treatment response, and future prognosis.

DETAILED DESCRIPTION:
"Idiopathic gastroparesis" is a poor term to describe this very heterogeneous syndrome. Pathophysiology may not be "idiopathic," but merely unidentifiable with conventional methods suggested for gastroparesis. The diagnosis of "gastroparesis" suggests that delayed gastric emptying is the underlying cause of symptoms, but this description fails to explain the variable presentation. There are fundamental differences in pathophysiology, clinical presentation, severity, and future prognosis among patients with idiopathic gastroparesis. Understanding these differences is necessary in order to provide cost-effective treatment in these patients.

We believe our clinical classification for gastroparesis is a clinical useful tool in the management of patients with idiopathic gastroparesis to predict clinical severity, treatment response, and future prognosis. Patients with vomiting-predominant gastroparesis will be more likely to have an underlying cause, such as viral infection or impaired glucose tolerance with vagal neuropathy. Their symptoms will likely be persistent. Patients with dyspepsia-predominant gastroparesis mimic those with functional dyspepsia and are unlikely to have complications such as weight loss, and dehydration. The necessity of enteric feeding in these patients is also unlikely. Prokinetics may help since delayed gastric emptying may contribute to epigastric pain or postprandial distress. Finding and treating small intestinal bacterial overgrowth as well as suggesting lifestyle and dietary modifications may be helpful. Patients with regurgitation-predominant gastroparesis may benefit most by improving their delayed gastric emptying. Their gastroparesis may cause reflux-like symptoms, especially at night.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of gastroparesis (nausea, vomiting, bloating, dyspepsia, early satiety, or effortless regurgitation) >1 month in duration.
* Abnormal 4-hour gastric emptying scan within the past 3 months.
* Initial investigation, based on the AGA Technical Review for gastroparesis, is non-diagnostic for an underlying cause

Exclusion Criteria:

* Presence of endocrine or metabolic diseases: type 1 or type 2 diabetes, hypothyroidism, renal failure, adrenal insufficiency.
* Presence of post-surgical gastroparesis: gastric surgery with vagotomy (with or without gastric resection, esophagectomy; surgery without vagotomy (fundoplication, bariatric surgery, heart-lung transplant).
* Presence of neuromuscular diseases: multiple sclerosis, chronic idiopathic demyelinating polyneuropathy, myotonic dystrophy.
* Presence of connective tissue diseases: systemic sclerosis, mixed connective tissue disorder, polymyositis, dermatomyositis, lupus.
* Presence of autonomic diseases: Central (Parkinson, multiple system atrophy, Lewy body disease, brainstem disease) or Peripheral (idiopathic dysautonomia, amyloidosis, immune-mediated disease, vitamin B12 deficiency, mitochondrial disorder, porphyria, hereditary sensory autonomic neuropathy).
* Presence of paraneoplastic syndrome: small cell lung cancer, multiple myeloma, breast cancer, lymphomas, pancreatic cancer.
* Taking dopamine agonists on a daily basis.
* Presence of known viral infection (Epstein-Barr, cytomegalovirus, herpes simplex, rotavirus), Chagas disease.
* Presence of gastric outlet, small bowel or colon mechanical obstruction.
* Presence of gastric electrical stimulator.
* Non-ambulatory patients: bed-ridden, nursing home resident, etc.
* Presence of active cancer or undergoing cancer treatment.
* Less than 16 years old.
* Pregnancy.
* Unable to provide informed consent.
* Prisoners.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects presenting to the University of Louisville Motility Center with newly diagnosis of idiopathic gastroparesis
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2010-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Incidence of poor outcome | 3 years
  Compare the incidence of any one of the following indicators of poor outcome between subjects with vomiting-predominant, dyspepsia-predominant, and regurgitation-predominant idiopathic gastroparesis:
  i) Developing new weight loss of >10% due to gastroparesis compare to weight at study baseline ii) Gastric failure (severe symptoms requiring G or J tube or TPN) iii) Death

SECONDARY OUTCOMES:
Clinical severity | 1 year
  Compare the prevalence of the pre-defined indicators of clinical severity between subjects with vomiting-predominant, dyspepsia-predominant, and regurgitation-predominant at study baseline.
Incidence of treatment success | 3 years
  Compare the incidence of pre-defined indicators of treatment success between the predominant-symptom subgroups.
Potential etiology of "idiopathic" gastroparesis | 1 year
  Compare the prevalence of pre-defined potential etiology between the predominant-symptom subgroups.
Prognostic indicators for idiopathic gastroparesis | 3 years
  Odd-ratios for developing the poor and good outcome during follow-up will be determined for pred-defined potential prognostic indictors obtained at the baseline visit.
Prevalence of obesity, metabolic syndrome and impaired glucose tolerance | 1 year
  Prevalence of obesity, metabolic syndrome and impaired glucose tolerance will be compared between the predominant-symptom subgroups and Subjects with and without gastroparesis complications.

CONTACTS AND LOCATIONS:
Overall Officials: John M. Wo, MD, Principal Investigator — University of Louisville School of Medicine
Locations (1):
- University of Louisville, Louisville, Kentucky, United States